CLINICAL TRIAL: NCT06449495
Title: Treatment of Balance and Coordination Disorders in the Pediatric Population With the Virtual Reality System Nirvana.
Brief Title: Virtual Reality for Pediatric Motor Rehabilitation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIP 1061
Record Dates: First submitted 2023-10-17; First posted 2024-06-10 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Coordination and Balance Disturbances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- coordination and balance disorders (Experimental): Subjects will undergo treatment with NIRVANA lasting 45 minutes for 5 sessions per week for 4 weeks combined with equal dose of task-oriented physiotherapy treatment.
  Interventions: Device: NIRVANA

INTERVENTIONS:
Device: NIRVANA — NIRVANA is a medical device using semi-immersive virtual reality for motor and cognitive neuro-rehabilitation.
  NIRVANA creates a "sensory room" where the patient can have an immersive and stimulating experience by interacting directly with different realistic scenarios. The system creates different scenarios on the wall or floor, and the patient interacts with the stimuli provided. A motion-analysis device detects the patient's behavior and based on the projected environment provides highly stimulating and rehabilitative audiovisual feedback with full whole-body immersion. The system is preconfigured with a series of exercises, which can be customized based on different types of patients, intervening on the level of difficulty, speed of execution and sensitive area of the projection.

SUMMARY:
Balance and coordination disorders limit the achievement of autonomy in movement and activities of daily living in pediatric population. There are several systems that can be used to treat balance and coordination disorders and those that use virtual reality, such as NIRVANA, are becoming increasingly popular. The primary objective of this post-market clinical investigation is to evaluate the efficacy of the semi-immersive virtual reality platform NIRVANA (BTS Bioengineering), in accordance with the protocol defined at IRCCS Medea in Bosisio Parini, in children with balance and coordination disorders on both motor function and cognitive processes that are indirectly stimulated.

DETAILED DESCRIPTION:
Balance and coordination disorders limit the achievement of autonomy in movement and activities of daily living.

Among the various conditions commonly associated with balance and gait deficits in the pediatric population, neurological diseases represent an important subgroup, as do neurodevelopmental disorders. Children with balance and coordination problems typically have difficulty walking independently and manifest a gait characterized by an enlarged base of support and are generally prone to frequent falls.

Coordination deficits also result in a reduction in the fluidity of functional gestures with a consequent negative impact on quality of life.

Not only that, in the presence of the above-mentioned problems, psycho-motor retardation is also often evident in children, consequently presenting cognitive, relational and learning problems as well.

There are several systems that can be used to treat balance and coordination disorders; in particular, those that use virtual reality systems such as NIRVANA are becoming increasingly popular. This device has been used in subjects with neurological disorders (Stroke, Parkinson's, and Multiple Sclerosis) with good results in both motor and visuocognitive areas. To date there are still few studies of this device in the pediatric setting, although its effectiveness in both autism spectrum disorders and global developmental delays is beginning to be explored.

The primary objective of this post-market clinical investigation is to evaluate the efficacy, in the context of its intended use, of the semi-immersive virtual reality platform NIRVANA (BTS Bioengineering), in accordance with the protocol defined at IRCCS Medea in Bosisio Parini, in children with balance and coordination disorders on both motor function and cognitive processes that are indirectly stimulated. Additional objective is to confirm the safety of the device, with the possibility of detecting any emerging risks with respect to expected performance. Secondary objective is to identify guidelines for use in clinical practice of the NIRVANA device with respect to pediatric populations undergoing treatment. Patients undergo a combined rehabilitation treatment consisting of 20 sessions with Nirvana and 20 sessions of physiotherapy (age >7aa) or psychomotor therapy (age <=7aa) over four weeks for a total of 40 sessions. The same subjects undergo clinical-functional assessments before and at the end of treatment:

* Stabilometry to assess balance with defined protocol on GAIT (BTS) platforms
* GMFM-88 o PBerg
* Continuous Performance Test (CPT or KCPT) sustained attention assessment test.

ELIGIBILITY:
Inclusion Criteria:

* balance or coordination disorders of different etiology: tumor, post-traumatic, neurodegenerative, syndromic, congenital, or associated with neurodevelopmental delay. - - - age between 4 and 17 years
* independent ambulation
* ability to understand simple verbal instructions.

Exclusion Criteria:

* adult
* wheelchair-bound
* major cognitive and behavioural problems.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2012-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Stabilometry with force platforms | T0(pre-training),T1 (after 4 weeks of training)
  Evaluation of static balance
Gross Motor Function Measure-88 (GMFM-88) | T0(pre-training),T1 (after 4 weeks of training)
  Evaluation of the motricity
Pediatric Berg Balance Scale (PBBS) | T0(pre-training),T1 (after 4 weeks of training)
  Functional balance

SECONDARY OUTCOMES:
Continuous Performance Test (CPT or KCPT) | T0(pre-training),T1 (after 4 weeks of training)
  Test for substained attention

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Irccs Eugenio Medea, Bosisio Parini, Lecco
  - Irccs Eugenio Medea, Conegliano, Treviso
  - Associazione "La Nostra Famiglia" - Polo Ospedaliero di Neuroriabilitazione, Piazza Di Summa presso ex Complesso Ospedaliero Regionale "A. Di Summa", Brindisi